CLINICAL TRIAL: NCT05381844
Title: Quantification of Antisense VIH-1 Transcripts and Comparison in Different Groups of Patients
Brief Title: Quantification of Antisense HIV RNA in Patients
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C21-16; 2021-A02266-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: HIV-1-infection
Keywords: HIV-1
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells obtained from a 30 ml EDTA blood sample. PBMCs will be frozen at -80°C before analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV-1-infected, untreated: Patients recently diagnosed with chronic HIV-1-infection with detectable HIV-1 RNA in plasma, sampled before treatment initiation
  Interventions: Other: Blood sampling
- HIV-1-infected, undetectable viral load: Patients with chronic HIV-1 infection on antiretroviral treatment for less than a year, with a plasma HIV-1 RNA < 50 copies/ml plasma since at least 6 months
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 30 ml blood sampling for virological research

SUMMARY:
The objective of this study is to quantify the expression levels of the HIV-1 unspliced sense transcript and of total HIV-1 antisense transcripts in PBMCs of HIV-1-infected persons, either still untreated or virologically controlled on treatment, and to investigate their correlations with the HIV reservoir as assessed by the quantification of total and integrated HIV-1 DNA.

DETAILED DESCRIPTION:
The research team will quantify the expression level of total HIV-1 antisense transcripts in PBMCs from two groups of HIV-1-infected persons: still untreated and virologically controllled on treatment.

The research team will also study (i) the correlation between the expression level of total HIV-1 antisense transcripts and the levels of total and integrated HIV-1 DNA in PBMCs, (ii) the correlation between the expression level of the unspliced HIV-1 sense transcript and the levels of total and integrated HIV-1 DNA in PBMCs, (iii) the correlation between the expression levels of total HIV-1 antisense transcripts and the level of the unspliced HIV-1 sense transcript in PBMCs, (iv) whether the correlations are different in the two groups of HIV-1-infected persons : still untreated patients vs. patients with virological control on antiretroviral treatment. Quantification of viral transcripts will rely on quantitative RT-PCRs, yielding the quantity of viral RNAs, normalized on the expression of 2 housekeeping genes, and on a digital RT-PCR, yielding the absolute number of viral RNA copies.

The quantification of total and integrated HIV-1 DNA will rely on a quantitative PCR yielding the number of HIV-1 DNA copies/million of PBMCs, according to the technique described in Tremeaux P et al, EBioMedicine 2019;41:455-64. The percentage of intact proviral DNA will be estimated according to the technique described in Bruner KM et al, Nature 2019; 566 :120-5

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* ability to understand the objectives and protocols of the research and to sign the informed consent

  * group 1 : treatment-naive patients with a detectable HIV-1 viral load
* Have not received any antiretroviral treatment
* At the chronic stage as determined during the clinical examination and confirmed by a western blot complete HIV antigens ("env" bands (gp 120 and 160). + "gag" and "pol" bands) with the presence of p31+

  *Group 2: patients with chronic HIV-1 infection on antiretroviral therapy efficient
* Have been on antiretroviral therapy for less than a year
* With a plasma HIV RNA < 50 copies/mL of blood for at least 6 months

Exclusion Criteria:

* ongoing HIV primary infection
* coinfection with HIV-2 or HTLV-1/2
* ongoing AIDS-defining clinical condition
* ongoing infectious disease of any type
* ongoing immunosuppressive treatment
* incompetent adults, persons under the protection of a conservator, tutor or guardian
* participation in a trial testing a medication in the 3 months preceding blood sampling
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected adults, before treatment, or with undetectable viral load on treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
HIV-1 antisense transcripts in PBMCs | 30 months
  Quantification of total antisense transcripts with quantitative PCR and digital RT-PCR

SECONDARY OUTCOMES:
Correlation between HIV-1 antisense transcripts and HIV-1 DNA in PBMCs | 30 months
  Study of the correlation between the expression level of total HIV-1 antisense transcripts and the level of total and integrated HIV-1 DNA in PBMCs
Correlation between unspliced HIV-1 sense transcripts and HIV-1 DNA in PBMCs | 30 months
  Study of the correlation between the expression level of unspliced HIV-1 sense transcripts and the level of total or integrated HIV-1 DNA in PBMCs
Correlation between HIV-1 sense and antisense transcripts in PBMCs | 30 months
  Study of the the correlation between the expression level of total HIV-1 antisense transcripts and the level of unspliced HIV-1 sense transcripts in PBMCs
Comparison of untreated patients vs. patients with virological control on treatment. | 30 months
  Study whether the correlations are different in HIV-1-infected persons with ongoing viral replication and persons with virological control on antiretroviral treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-Paul VIARD, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tremeaux P, Lenfant T, Boufassa F, Essat A, Melard A, Gousset M, Delelis O, Viard JP, Bary M, Goujard C, Rouzioux C, Meyer L, Avettand-Fenoel V; ANRS-SEROCO and PRIMO cohorts. Increasing contribution of integrated forms to total HIV DNA in blood during HIV disease progression from primary infection. EBioMedicine. 2019 Mar;41:455-464. doi: 10.1016/j.ebiom.2019.02.016. Epub 2019 Feb 23. PMID 30803934
- [Background] Bruner KM, Wang Z, Simonetti FR, Bender AM, Kwon KJ, Sengupta S, Fray EJ, Beg SA, Antar AAR, Jenike KM, Bertagnolli LN, Capoferri AA, Kufera JT, Timmons A, Nobles C, Gregg J, Wada N, Ho YC, Zhang H, Margolick JB, Blankson JN, Deeks SG, Bushman FD, Siliciano JD, Laird GM, Siliciano RF. A quantitative approach for measuring the reservoir of latent HIV-1 proviruses. Nature. 2019 Feb;566(7742):120-125. doi: 10.1038/s41586-019-0898-8. Epub 2019 Jan 30. PMID 30700913